CLINICAL TRIAL: NCT02568917
Title: Effectiveness of Atraumatic Restorative Treatment and Conventional Restorations in Primary and Permanent Dentition: A Practice-based Clinical Trial
Brief Title: Effectiveness of ART and Conventional Treatment - Practice-based Clinical Trial
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: There was a problem with the municipality and they have choose to suspend it.
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Daniela Prócida Raggio, Associated Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EFFART
Record Dates: First submitted 2015-09-29; First posted 2015-10-06 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Dental Caries
Keywords: Dental Atraumatic Restorative Treatment; Composite Resins; Primary Teeth; Permanent Teeth; Clinical Effectiveness; Cost Analysis
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Restoration (Active Comparator): Conventional Restoration - Composite Resin (Bulk Fill)
  Interventions: Procedure: Conventional Restoration - Composite Resin (Bulk Fill)
- Atraumatic Restorative Treatment (Experimental): Atraumatic Restorative Treatment - Ketac Molar Easy Mix
  Interventions: Procedure: Atraumatic Restorative Treatment - Ketac Molar Easy Mix

INTERVENTIONS:
Procedure: Atraumatic Restorative Treatment - Ketac Molar Easy Mix — Occlusal and occlusal-proximal ART restorations in primary and permanent molars using the high viscosity GIC Ketac Molar Easy mix will be performed. No local anesthesia will be used. Infected carious tissue will be removed with hand instruments, and the cavities restored with GIC (Glass Ionomer Cement). The cavity will be filled with GIC. After the press-finger technique, the excess of material will be removed and occlusion will be checked.
  Arms: Atraumatic Restorative Treatment
Procedure: Conventional Restoration - Composite Resin (Bulk Fill) — Occlusal and occlusal-proximal composite resin restorations in primary and permanent molars using the Scotchbond Multi-purpose adhesive system and the Filtek Bulk Fill composite resin wil be performed. Local anesthesia can be used if necessary. Access to caries lesion will be done using a round bur. Infected carious tissue will be removed with hand instruments. The cavity will be etched for 15 seconds followed by rising and drying for the same amount of time. The cavity will be restored with composite resin. Occlusion will be checked.
  Arms: Conventional Restoration

SUMMARY:
Background: Dental caries is still a public health problem among Brazilian children and doubts still exist regarding the most effective restorative technique. The aim of this pragmatic randomized clinical trial is to evaluate the effectiveness of single and multiple-surfaces restorations performed following the Atraumatic Restorative Treatment (ART) premises compared with Conventional Treatment (CT) in primary and permanent teeth.

Methods: A total of 1,214 5-to-13 years-old children with at least one single or multiple-surface dentin caries lesion in primary or permanent molars will be selected in the public schools of Barueri-SP. The participants will be randomly divided into 2 groups: CT (Filtek Bulk Fill - 3M) and ART (Ketac Molar Easy Mix - 3M) and treated by ten untrained dentists in a dental office inside the schools. The restorations will be evaluated after 6, 12 and 24 months by an independent trained and calibrated examiner. The restoration and tooth survival, the cost-effectiveness analysis between the two groups and the operator preference of the treatment regarding the techniques will be also evaluated. Kaplan-Meier survival analysis and log-rank test will be applied to the survival of restorations. All the average event rates in the two groups will be modelled and compared with a Cox proportional hazard shared frailty model since there is an operator cluster-effect. The significance level for all analyses will be 5%.

DETAILED DESCRIPTION:
Background: Dental caries is still a public health problem among Brazilian children and doubts still exist regarding the most effective restorative technique. The aim of this pragmatic randomized clinical trial is to evaluate the effectiveness of single and multiple-surfaces restorations performed following the Atraumatic Restorative Treatment (ART) premises compared with Conventional Treatment (CT) in primary and permanent teeth.

Methods: A total of 1,214 5-to-13 years-old children with at least one single or multiple-surface dentin caries lesion in primary or permanent molars will be selected in the public schools of Barueri-SP. The participants will be randomly divided into 2 groups: CT (Filtek Bulk Fill - 3M) and ART (Ketac Molar Easy Mix - 3M) and treated by ten untrained dentists in a dental office inside the schools. The restorations will be evaluated after 6, 12 and 24 months by an independent trained and calibrated examiner. The restoration and tooth survival, the cost-effectiveness analysis between the two groups and the operator preference of the treatment regarding the techniques will be also evaluated. Kaplan-Meier survival analysis and log-rank test will be applied to the survival of restorations. All the average event rates in the two groups will be modelled and compared with a Cox proportional hazard shared frailty model since there is an operator cluster-effect. The significance level for all analyses will be 5%.

Discussion: Our hypothesis is that despite similar expected effectiveness between ART using high viscosity GIC and conventional treatment using composite resin when treating single or multiple-surface in posterior primary and permanent teeth, ART presents superior cost-effectiveness. The results of this trial will support decision-making by clinicians and policy makers

Keywords: atraumatic restorative treatment, composite resin, glass ionomer cement, randomized clinical trial, cost effectiveness analysis

ELIGIBILITY:
Inclusion Criteria:

* Children aging between 6 and 14 years
* presenting good health conditions
* spontaneous demand for treatment by parents or legal guardians
* whose parents or legal guardians accept and sign the consent form
* with at least one occlusal or occlusal proximal caries lesion in primary or permanent molars
* only occlusal and/or occlusal-proximal surfaces with caries lesions with dentin involvement

Exclusion Criteria:

* severe behavioral issues
* presence of fistula or abscess near the selected tooth
* presence of pulp exposure in the selected tooth
* presence of mobility in the selected tooth

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
The restoration survival | Every 6 months up to 18 months
  The treatments will be classified as successful when they present a clinical satisfactory aspect. Otherwise, "minor failures" will be analyzed. "Minor failures" are those in which there is a defect in the restoration/crown, but it does not interfere with the tooth health.

SECONDARY OUTCOMES:
Longevity of the tooth | Every 6 months up to 18 months
  For evaluation of this outcome will be considered "successful" the restoration even a minor failure of the restoration (scores 00 to 30). Only the restored teeth that presents symptoms of pulp inflammation or need for extraction (scores 40 and 50) will be considered as "failure", since it cannot be considered as a successful treatment for the tooth.
  The main objective of a restoration is to aprovide patient a condition for improved hygiene, can enable inactivation of injury, plus the return of the masticatory function of that tooth, so the scores considered "minor failures" is not considered failure for the tooth (Bonifácio et al., 2012).
Cost-effectiveness assessment | Through study completion, an average of 18 months
  Treatment costs will be calculated considering professional costs and procedure costs. In order to calculate the professional cost the time spent in each session will be converted in hours and multiplied by the medium income of the dentist per hour as related by the Brazilian Ministry of Labour and Employment ($36,23). On the other hand, to estimate the procedure cost, it will be considered both variable cost, which includes electricity and equipment depreciation, and materials cost. To calculate the equipment depreciation (peripherals, dental chair and instrumental), we will consider their price, the lifespan of five years and a monthly use of 160 hours, using an estimate value per hour of $1,81. All materials used in each procedure will have their specifications and quantity registered. Prices will be inferences from the market value converted in US Dollars and obtained by the medium of the values from different places that commercialized the referred products.

OTHER OUTCOMES:
Preference of the treatments by dentists | Baseline and after 6 months
  The preference for one of the treatments performed by the dentist will be evaluated at the end of the operative phase of the study. Thus, we aimed to identify which is the preferred procedure by professionals. To evaluate this outcome, a questionnaire composed of six items will be applied.
  This questionnaire was adapted from the study of Pani et al. (2014), which evaluated the preference of students with respect to composite and silver amalgam. The questionnaire was translated from English to Portuguese by a Brazilian dentist who is fluent in both languages (Appendix ) and adapted for comparing the composite resin and the atraumatic restorative treatment (use of glass ionomer cement). This questionnaire will be administered before and after the research in the participating dentists (operators).

CONTACTS AND LOCATIONS:
Overall Officials: Daniela P Raggio, Professor, Principal Investigator — University of Sao Paulo; Isabel C Olegário, PhD Student, Principal Investigator — University of Sao Paulo
Locations (1):
- University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olegario IC, Hesse D, Bonecker M, Imparato JC, Braga MM, Mendes FM, Raggio DP. Effectiveness of conventional treatment using bulk-fill composite resin versus Atraumatic Restorative Treatments in primary and permanent dentition: a pragmatic randomized clinical trial. BMC Oral Health. 2016 Aug 2;17(1):34. doi: 10.1186/s12903-016-0260-6. PMID 27485432